CLINICAL TRIAL: NCT02837445
Title: Clinical Evaluation of Safety and Effectiveness of the BackBeat Medical Moderato System in Patients With Hypertension: A Double-Blind Randomized Trial
Brief Title: Moderato System: A Double-Blind Randomized Trial Ver 1.1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BackBeat Medical Inc (Industry)
Collaborators: Massachusetts General Hospital (Other); MLM Medical Labs GmbH (Industry); nabios GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS-03 Ver 1.1
Record Dates: First submitted 2016-07-08; First posted 2016-07-19 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Hypertension Resistant to Conventional Therapy; Bradycardia; Atrioventricular Block
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Bradycardia; Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Eligible patients randomized after optimization phase to PHC ON for 6 months Patients continue standard or modified anti-hypertension medical regime at discretion of the investigator
  Interventions: Device: PHC ON
- Control (Placebo Comparator): Eligible patients randomized after optimization phase to pacemaker only (PHC OFF) for 6 months. Patients continue standard or modified anti-hypertension medical regime at discretion of the investigator
  Interventions: Device: PHC OFF

INTERVENTIONS:
Device: PHC ON — Eligible patients randomized after optimization phase to PHC ON for 6 months. Patients continue standard or modified anti-hypertension medical regime at discretion of the investigator
  Arms: Treatment
Device: PHC OFF — Eligible patients randomized after optimization phase to PHC OFF for 6 months. Patients continue standard or modified anti-hypertension medical regime at discretion of the investigator.
  Arms: Control

SUMMARY:
The purpose of this double blind randomized study is the evaluation of the safety and efficacy of the Moderato System.

The Moderato implantable pulse generator is indicated for patients who have hypertension and also require a dual chamber pacemaker in order to reduce their blood pressure.

The primary objectives of this study are to provide evidence of safety and clinical efficacy of the anti-hypertensive effects of the Moderato System. This will be accomplished by evaluating changes in blood pressure in an active treatment vs. a control patient population for a period of 6 months.

The device will be considered to have a clinical effectiveness with regard to its anti-hypertension functions if there is a statistically significant and clinically meaningful reduction in mean 24-hour ambulatory systolic blood pressure in the treatment group compared to the control group.

DETAILED DESCRIPTION:
Protocol CS-03 Ver 1.1 (NCT02837445) was amended at the advice of the Scientific Advisory to protocol CS-03 Version 3.0 with more stringent hypertension inclusion criteria and different observation intervals for efficacy and safety.

In CS-03 Version 3.0 the time of the primary efficacy endpoint was reduced from 6 months to 3 months post randomization which was deemed a suitable interval for the chronic effect, whereas for the safety endpoint, the period was lengthened from 6 month to 12 months post randomization to better monitor potential risks of the treatment on cardiac function (Blinding period was increased from 6 to 12 months). Protocols were thus split in order to allow better clarification to the difference in the time to the primary endpoints for efficacy and safety between the two CIP versions and simplify data analysis.

Protocol Ver 3.0 prescribes data analysis of all patients randomized under version 1.1 to be performed once they complete the 6 months follow-up as set in protocol version 1.1 (NCT0283744). It is expected that ~40 patients will be randomized according to protocol version 1.1 prior to the enrollment of patients according to protocol version 3.0. The results will be considered as interim analysis.

The recruitment for the protocol version 1.1 is now completed. Total of 47 patients were randomized according to protocol version 1.1 and all patients completed the follow-up period for the primary endpoint.

Patients are currently being followed up for the study "extension period".

ELIGIBILITY:
Inclusion Criteria:

* Subject requires an implant or replacement a of dual chamber pacemaker
* Stable (at least one month) hypertension treatment with at least 1 anti-hypertensive drug, which is anticipated to be maintained for 7 months.
* Average day time (7AM-10PM) ambulatory systolic blood pressure ≥ 130 mmHg and office blood pressure ≥140 mmHg.
* Subject lives in the proximity of the study center, which permits compliance with study visits for at least 7 months.

Exclusion Criteria:

* Known secondary cause of HTN.
* Average ambulatory or office systolic BP > 195 mmHg.
* Permanent atrial fibrillation.
* History of significant paroxysmal atrial fibrillation/flutter burden (defined as >25% of beats).
* Cardiac ejection fraction <50%.
* Symptoms of heart failure, NYHA Class II or greater.
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy or inter-ventricular septal thickness ≥ 15 mm.
* Subject is on dialysis.
* Subject has an estimated Glomerular Filtration Rate < 30 ml/min/1.73 m²
* Prior neurological events (stroke or TIA) within the past year or events at a prior time that has resulted in residual neurologic deficit.
* Carotid artery disease.
* Known autonomic dysfunction.
* History of clinically significant untreated ventricular tachyarrhythmia or has experienced sudden death.
* Previous active device-based treatment for HTN.
* Existing implant, other than a pacemaker that needs replacing.
* Subject is or has the possibility of becoming pregnant and is unwilling of contraception during the study.
* Subject is unwilling or cannot provide Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2016-07-12 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Rate of composite of major cardiac events | 6 months post Randomization
  including heart failure, clinically significant arrhythmias eg, persistent or increased atrial fibrillation, serious ventricular arrhythmias, myocardial infarction, stroke, heart failure, renal failure and/or related safety events that result in death
Change in average 24 hour systolic ambulatory blood pressure | Week 3 pre Randomization and 6 months post Randomization

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof. MD, Principal Investigator — Asklepios Klinik St. Georg
Locations (12):
- Austria (2):
  - Krankenhaus der Elisabethinen, Linz
  - Medical University Vienna, Vienna
- UZ Brussel - Heart Rhythm Management Center, Brussels, Belgium
- Na Homolce Hospital, Prague, Czechia
- Semmelweis University Heart and Vascular Center, Budapest, Hungary
- P. Stradins Clinical University Hospital, Riga, Latvia
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania
- Poland (5):
  - Medical University of Gdansk, Gdansk
  - Szpital Kliniczny Przemiemienia Panskiego, Poznan
  - Pomeranian Medical University Hospital no. 2, Szczecin
  - Samodzielnym Publicznym Centralnym Szpitalem Klinicznym, Warsaw
  - Silesian Center for Heart Diseases, Zabrze

REFERENCES:
- [Derived] Chovanec M, Merkely B, Sokal A, Petru J, Kralovec S, Drtina T, Mudroch M, Geller L, Osztheimer I, Morawski S, Mika YH, Fischer A, Evans SJ, Aviv R, Rosenthal N, Burkhoff D, Kuck KH, Neuzil P. Pressure-Volume Analysis Demonstrates Short- and Long-Term Hemodynamic Effects of Atrioventricular Interval Modulation Therapy in Hypertension. JACC Clin Electrophysiol. 2025 Nov;11(11):2493-2504. doi: 10.1016/j.jacep.2025.06.017. Epub 2025 Aug 13. PMID 40801869
- [Derived] Kalarus Z, Merkely B, Neuzil P, Grabowski M, Mitkowski P, Marinskis G, Erglis A, Kazmierczak J, Sturmberger T, Sokal A, Pluta S, Geller L, Osztheimer I, Malek F, Kolodzinska A, Mika Y, Evans SJ, Hastings HM, Burkhoff D, Kuck KH. Pacemaker-Based Cardiac Neuromodulation Therapy in Patients With Hypertension: A Pilot Study. J Am Heart Assoc. 2021 Aug 17;10(16):e020492. doi: 10.1161/JAHA.120.020492. Epub 2021 Aug 13. PMID 34387126